CLINICAL TRIAL: NCT06863402
Title: Nemtabrutinib and Pembrolizumab in Patients With Richter Transformation: A Phase II Study
Brief Title: Nemtabrutinib and Pembrolizumab for the Treatment of Richter Transformation, Diffuse Large B-cell Lymphoma Subtype
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-3586924; NCI-2025-01256 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3586924 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2025-02-26; First posted 2025-03-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Richter Syndrome; Diffuse Large B-Cell Lymphoma; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Specimen Handling; Biopsy; ARQ531; pembrolizumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (nemtabrutinib, pembrolizumab) (Experimental): Patients receive nemtabrutinib PO QD on days 1-21 of each cycle and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients undergo ECHO or MUGA during screening, PET/CT or CT and blood sample collection throughout the trial. Patients may also undergo bone marrow biopsy throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: Multigated Acquisition Scan; Drug: Nemtabrutinib; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo ECHO
  Other Names: EC
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Nemtabrutinib — Given PO
  Other Names: ARQ 531; ARQ-531; ARQ531; Bruton's Tyrosine Kinase Inhibitor ARQ 531; BTK Inhibitor ARQ 531; MK-1026
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; QL2107; RPH 075; RPH-075; RPH075; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well nemtabrutinib in combination with pembrolizumab works in treating patients with Richter transformation, diffuse large B-cell lymphoma subtype (RT-DLBCL). Nemtabrutinib is in a class of medications called kinase inhibitors. It blocks a protein called BTK, which is present on B-cells (a type of white blood cell) in cancers such as Richter transformation at abnormal levels. This may help keep cancer cells from growing and spreading. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Giving nemtabrutinib in combination with pembrolizumab may kill more cancer cells in patients with RT-DLBCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the preliminary efficacy of nemtabrutinib and pembrolizumab as measured by the overall response rate (ORR) after 6 cycles for enrolled patients with Richter transformation, diffuse large B-cell lymphoma subtype (RT-DLBCL).

SECONDARY OBJECTIVES:

I. To further evaluate preliminary efficacy as measured by complete response rate (CRR), duration of response (DOR), progression-free survival (PFS), and overall survival (OS) for enrolled patients.

II. To evaluate the safety and tolerability of nemtabrutinib and pembrolizumab combination treatment for RT-DLBCL.

III. Evaluate patient-reported outcomes on quality of life and disease-related symptoms and side-effects.

EXPLORATORY OBJECTIVES:

I. To investigate the effects of nemtabrutinib and pembrolizumab exposure on peripheral blood mononuclear cell (PBMC) composition, particularly T-regulatory and cytotoxic T/natural killer (NK)-cell populations and correlate with clinical outcome/response.

II. To investigate the impact of nemtabrutinib and pembrolizumab on the fitness, function, and "stem-like" properties of chimeric antigen receptor (CAR) T-cells manufactured from specimens both pre- and post-treatment.

III. To evaluate the potential late effects of this novel combination treatment on CAR T-cell therapy and/or allogeneic hematopoietic stem cell transplant treated patients.

IV. To evaluate molecular subtypes of RT-DLBCL using multiomic and probabilistic classification approaches, as well as tumor characteristics (e.g. mutational profile and total mutational burden, PD-L1 expression, etc.), and correlate with clinical outcomes for enrolled subjects.

V. To evaluate pharmacokinetic (PK) and pharmacodynamic (PD) data obtained from analyses of blood specimens collected throughout treatment (for both Nemtabrutinib as well as Pembrolizumab) to enable PopPK modeling, exposure-response analyses, and integrated assessments of PK/PD data with safety, efficacy, and activity.

OUTLINE:

Patients receive nemtabrutinib orally (PO) once daily (QD) on days 1-21 of each cycle and pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 35 cycles (2 years) in the absence of disease progression or unacceptable toxicity. Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) during screening, positron emission tomography (PET)/computed tomography (CT) or CT and blood sample collection throughout the trial. Patients may also undergo bone marrow biopsy throughout the trial.

After completion of study treatment, patients are followed up at 30 days then every 6 months for 3 years after completion of therapy or until death, whichever comes first, for a total of up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven Richter transformation, diffuse large B-cell lymphoma subtype (RT-DLBCL) from an antecedent or concurrently diagnosed chronic lymphocytic leukemia (CLL) and/or small lymphocytic lymphoma (SLL).
* Be ineligible for frontline anthracycline-based chemoimmunotherapy (determined by treating investigator) OR have clinical evidence of disease progression after any prior treatment for RT-DLBCL.
* Participants who have adverse events (AEs) due to previous anti-cancer therapies must have recovered to ≤ grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤ grade 2 neuropathy are eligible.

  * Note: Participants who have lingering cytopenias from prior anti-cancer therapy or progressive disease may be eligible at the discretion of the study principal investigator (PI), provided they meet all other study criteria.
* Have measurable disease as determined by imaging (by positron-emission tomography [PET] and/or computed tomography [CT] scans), immunohistochemistry, and/or flow cytometry, as per the Cheson criteria.
* Have the ability to swallow and retain oral medication.
* Age 18 years and older on the day of signing informed consent.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Be free from other malignancy within 2 years prior to enrollment (with the exception of CLL/SLL, low-risk and early stage [T1-T2a- Gleason score ≤ 6, and prostate-specific antigen [PSA] < 10 ng/mL] prostate cancer, or localized skin cancer that has undergone potentially curative therapy).
* Absolute neutrophil count: ANC ≥ 500 cells/µL (without G-CSF dose within the last 7 days prior to initiation of study treatment
* Platelets: ≥ 25,000/µL -not requiring transfusion within the last 3 days prior to initiation of study treatment). Patients on medications that increase bleeding risk (e.g. systemic anticoagulation, anti-platelet therapies, etc.) must have a platelet count ≥50,000 /µL and have no history of major bleeding.
* Hemoglobin: ≥ 7gm/dL (transfusion support allowed).
* Total bilirubin: ≤ 1.5 x upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 x ULN.
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase [SGPT]): ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastases).
* Creatinine clearance (CrCl): ≥ 30 mL/min (per Cockroft-Gault equation).
* International normalized ratio (INR) (prothrombin [PT]/activated partial thromboplastin time [aPTT]): ≤ 1.5 x ULN, unless participant is receiving anticoagulant therapy, as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
* Patients with history of human immunodeficiency virus (HIV) infection are potentially eligible (after conferring with the PI) if they meet ALL of the following criteria:

  * Must have a CD4+ T-cell count ≥ 350 cells/mm^3 AND an HIV viral load below the detectable level as per locally available testing at the time of screening
  * It is advised that participants must not have had any AIDS-defining opportunistic infections within the past 12 months.
  * Participants on anti-retroviral therapy (ART) must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (day 1) and agree to continue ART throughout the study.
  * The combination ART regimen must not contain any antiretroviral medications that interact with strong CYP3A4 inhibitors/inducers/substrates (<https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers>). Participants receiving ART that are strong CYP3A4 inducers are not eligible to be included in the study.
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to randomization.

Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention. Hepatitis B screening tests, including HBsAg and hepatitis B core antibodies (anti-HBc), are required for all participants.

* Participants with history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening (Participants must have completed curative anti-viral therapy at least 4 weeks prior to the first administration of the study treatment).
* A person of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Participants of child-bearing potential must agree to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Should a person of child-bearing potential become pregnant or suspect they are pregnant while they or their partner is participating in this study, they should inform their treating physician immediately.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137).
* Has received prior systemic anti-cancer therapy within 5 half-lives of last dose (or within 30 days for cellular therapy or investigational agents, or within 100 days post allogeneic hematopoietic stem cell transplantation and without any grade ≥ 2 graft versus host disease) prior to enrollment.
* Has received prior radiotherapy within 2 weeks of start of study intervention or has radiation related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-central nervous system (CNS) disease is permitted. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study intervention.
* Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed or messenger ribonucleic acid (mRNA) vaccines is allowed.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (daily dose exceeding 10 mg of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 2 years.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention. Has severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients.
* Has severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid allowed).
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has not adequately recovered from major surgery or has ongoing surgical complications.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Patients with pathologically confirmed Hodgkin-like RT (RT-classical Hodgkin's lymphoma [cHL]).
* Estimated life expectancy of < 1 month as determined by the treating investigator.
* Uncontrolled active illness including but not limited to heart failure, unstable ischemic heart disease, arrhythmia, psychiatric illness, acute renal failure, and any other conditions that would reasonably be expected to limit compliance with the study protocol.
* Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV deoxyribonucleic acid [DNA]) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.
* Corrected QT interval (QTc) prolongation (defined as a Fridericia's corrected QT [QTcF] > 450 msecs) or other significant electrocardiogram (ECG) abnormalities including second degree atrioventricular (AV) block type II, third degree AV block, or bradycardia (ventricular rate less than 50 beats/min).
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Unwilling or unable to follow protocol requirements.
* Received any other investigational agent within 30 days prior to enrollment.
* HIV-infected participants with a history of Kaposi's sarcoma and/or multicentric Castleman's disease.
* History of severe bleeding disorder defined as an ongoing congenital or acquired condition that leads to an increased likelihood of bleeding.NOTE: Patients on active anti-coagulation, anti-platelet therapies, and other medications that may increase bleeding risks may be allowed on study, permitted that these potentially interacting drugs may be safely held in the setting of thrombocytopenia, and at the discretion of the treating investigator and with close monitoring.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has had an allogeneic tissue/solid organ transplant. Note: Patients with prior allogeneic hematopoietic stem cell transplant or allogeneic cellular therapy are allowed, provided they meet they meet the washout period.
* Use of medications that are strong CYP3A4 inhibitors or inducers or P-gp and/or BCRP substrates with a narrow therapeutic index within 14 days prior to first dose of study treatment or 5 half-lives of the given drug, whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | After 6 cycles (approximately 18 weeks) (1 cycle = 21 days)
  Will be defined as having either a complete response (CR) or partial response (PR) as per Cheson et al., 2014. Will be summarized using frequencies and relative frequencies.
Quality of life | Up to 3 years after completion of study treatment
  Tolerability and patient-reported outcomes (PROs) assessed using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (version 3) . EORTC-C 30 is measure from nat at all (better) to very much (worse)
Quality of life -PRO CTCAE | Up to 3 years after completion of study treatment
  Will be evaluated using the patient reported outcome PRO CTCAE measurement system. Responses are scored on a 0-5 point scale where higher outcomes indicate worse

SECONDARY OUTCOMES:
Response outcomes | Up to 3 years after completion of study treatment
  CR, PR, stable disease (SD), CR+PR, and CR+PR+SD will be summarized using frequencies and relative frequencies, with response rates estimated using 90% credible regions obtained by Jeffrey's prior method.
Duration of response | From first PR (or greater) until disease progression or last follow-up, assessed up to 3 years after completion of study treatment
  Will be summarized using standard Kaplan-Meier methods, where the median will be estimated with a 90% confidence interval.
Overall survival | From treatment initiation until death due to any cause or last follow-up, assessed up to 3 years after completion of study treatment
  Will be summarized using standard Kaplan-Meier methods, where the medians will be estimated with 90% confidence intervals.
Progression-free survival | From treatment initiation until disease progression, death due to any cause, subsequent treatment, or last follow-up, assessed up to 3 years
  Will be summarized using standard Kaplan-Meier methods, where the medians will be estimated with 90% confidence intervals.
Incidence of adverse events | Up to 30 days after the last dose of study treatment
  Toxicities and adverse events will be reported using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be summarized by attribution and grade using frequencies and relative frequencies.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Cortese, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States